CLINICAL TRIAL: NCT05992038
Title: A Randomized Controlled Trial of AttraX® Putty vs. Conventional Open-wedge Osteotomy Without Gap Filler in Open-wedge Osteotomy
Brief Title: Use of a Putty as Gap Filler in Open-wedge Osteotomy
Acronym: AXOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, R.J.H. Custers, Principal investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 84534
Record Dates: First submitted 2023-07-26; First posted 2023-08-15 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteotomy; Gap filler; Postoperative pain; Randomized controlled trial; AttraX Putty
MeSH Terms: conditions — Pain, Postoperative | interventions — Osteotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Putty (Experimental): The osteotomy gap will be filled with a synthetic ceramic material, Putty
  Interventions: Procedure: Osteotomy with putty
- Conventional (Placebo Comparator): Osteotomy performed according to the conventional method, without gap filler
  Interventions: Procedure: Conventional osteotomy

INTERVENTIONS:
Procedure: Osteotomy with putty — Synthetic ceramic putty
  Arms: Putty
Procedure: Conventional osteotomy — conventional osteotomy
  Arms: Conventional

SUMMARY:
Rationale: Realignment osteotomies around the knee are a proven surgical treatment for unicompartmental knee osteoarthritis and a malalignment. Osteotomies can be very painful in the early postoperative phase. This is probably due to a combination of bony cut (bone pain) and postoperative hematoma (bleeding and leakage of the bone marrow) in the surrounding soft tissue. The AttraX® Putty can be used as a gap filler in open wedge osteotomies to potentially reduce postoperative pain by reducing the bleeding from the bone gap.

Objective: The main aim of this study is to determine whether early postoperative pain is decreased when the osteotomy gap is filled with AttraX® Putty, compared to conventional open wedge osteotomy without filling the gap. The secondary aims are faster accelerated rehabilitation/regaining function, reduction of local blood loss, accelerated bone union, comparable surgical accuracy, and the occurrence of (serious) adverse events.

Study design: Single-blinded, prospective, randomized controlled trial.

Study population: Adult patients qualifying for open-wedge tibial, open-wedge femur or double level osteotomy.

Intervention: According to a randomization scheme, the osteotomy gap will be filled with either the synthetic ceramic material AttraX® Putty or without a gap filler (conventional method).

Main study parameters/endpoints: The main study endpoint is the Numeric Rating Scale (NRS) pain during the first week postoperative. The secondary study endpoints are faster rehabilitation/regaining function, reduction of local blood loss, accelerated bone union, comparable surgical accuracy, and (serious) adverse events.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients may have the advantage of experiencing less pain postoperatively if they are treated with the AttraX® Putty, which can contribute to a faster rehabilitation. Risks to the AttraX® Putty group may include an allergic reaction, failure to promote bone fusion and excessive bone growth. However, the preclinical studies and clinical studies show that the use of AttraX® Putty is safe for use in humans.

DETAILED DESCRIPTION:
Rationale: Realignment osteotomies around the knee are a proven surgical treatment for unicompartmental knee osteoarthritis and a malalignment. Osteotomies can be very painful in the early postoperative phase. This is probably due to a combination of bony cut (bone pain) and postoperative hematoma (bleeding and leakage of the bone marrow) in the surrounding soft tissue. The AttraX® Putty can be used as a gap filler in open wedge osteotomies to potentially reduce postoperative pain by reducing the bleeding from the bone gap.

AttraX® Putty: AttraX® putty is a synthetic ceramic which consists of calcium phosphate granules and hydroxyapatite (ß-tricalcium phosphate (>90%)/hydroxyapatite(<10%)). It is Conformité Européenne (CE) marked as bone void filler and bone haemostasis implant. Unlike most other synthetic bone grafts which are only osteoconductive, AttraX Putty is both osteoconductive and osteoinductive. Moreover, AttraX® Putty could overcome the disadvantages of using autologous bone grafts and allografts, such as, donor site morbidity, increased surgical time, and disease transmission. Animal studies and a clinical study showed no difference in bone fusion between AttraX® Putty and autograft after instrumented thoracolumbar fusion.

Objectives: The main aim of this study is to determine whether early postoperative pain is decreased when the osteotomy gap is filled with AttraX® Putty, compared to conventional open wedge osteotomy without filling the gap. The secondary aims are faster accelerated rehabilitation/regaining function, reduction of local blood loss, accelerated bone union, comparable surgical accuracy, and the occurrence of (serious) adverse events.

Study design: Single-blinded, prospective, randomized controlled trial.

Study population: Adult patients qualifying for open-wedge tibial, open-wedge femur or double level osteotomy. A total of 40 patients will be included, 20 patients in the control group (without gap filler) and 20 patients in the AttraX Putty group (with AttraX® Putty as gap filler). Osteotomy in combinations with cartilage treatment and corrections above 10 mm will be excluded.

Main study parameters/endpoints: The main study endpoint is the Numeric Rating Scale (NRS) pain during the first week postoperative. The secondary study endpoints are the NRS pain during the second week, at 1 months, and at 3 months. Moreover, faster rehabilitation/regaining function, reduction of local blood loss, accelerated bone union, comparable surgical accuracy, and (serious) adverse events are secondary endpoints.

Study procedures: According to standard care, standing anteroposterior and lateral radiographs will be taken postoperatively during hospitalization. The subsequent follow-up moments will take place at the outpatient clinic. The follow-up moments take place at +1 month, +4 months, +6 months, and +1 year postoperatively at the outpatient clinic. The follow-up moment of +6 months is extra for this study. During this extra follow-up moment, a CT scan of the lower limb (+6 months postoperative) will be performed to be able to draw a conclusion about the bone union.

According to standard care, radiographs are performed at +1 day, +1 month, +4 months, and +1 year. An extra radiograph will be performed at +6 months. Using these radiographs, a conclusion can be drawn about the union rate and osteotomy accuracy.

Moreover, the preoperative and postoperative (+1 day) haemoglobin value will be analysed, according to standard care. Using the haemoglobin value one of the secondary outcomes can be determined (difference in haemoglobin value between preoperative and postoperative).

The rest of the data will be collected at -1 week, +1 day, +1 week, +2 weeks, +3 weeks, +1 months, + 3 months, +4 months, +6 months, and +1 year postoperatively. This will involve questionnaires (Knee Injury and Osteoarthritis Outcome Score (KOOS), EuroQol Five Dimensions Health Questionnaire (EQ-5D) and Kujala Patellofemoral Score), the NRS pain score, and measuring the calf or upper leg circumference. The calf or upper leg circumference is measured at the site where the open wedge osteotomy was performed. For a double-level osteotomy, it depends on where the open wedge osteotomy has taken place: the femur or the tibia. The location where the calf or upper leg circumference is to be measured will be marked with a marker. The patient will be given a tape measure to take home to measure the circumference in the morning. Using these data, the primary outcome and secondary outcomes can be answered.

If there is an indication for removal of the plate osteosynthesis (for example complaints of the plate after one year postoperative), the plate will be surgically removed, and a fine needle biopsy will be taken to analyse the newly formed bone. When indicated, the removal of the plate osteosynthesis will take place in the period from 12 months to 18 months postoperative.

Benefits and risks: Patients have the advantage of being checked more closely during follow-up. In addition, patients may have the advantage of experiencing less pain postoperatively if they are into the AttraX Putty group, which can contribute to an accelerated rehabilitation. Risks to the AttraX Putty group may include an allergic reaction, failure to promote bone fusion and excessive bone growth. However, the preclinical studies and clinical studies show that the use of AttraX® Putty is safe. Moreover, an extra CT scan and radiography are performed during this study. You will receive approximately 0.1 millisievert (mSv) of additional radiation because of this CT scan. By way of comparison: the 'ordinary' radiation that everyone in the Netherlands receives anyway is about ~2.9 mSv per year.

ELIGIBILITY:
Inclusion Criteria:

* indication for an open-wedge osteotomy of the femur, tibia or double level due to unicompartmental osteoarthritis (OA).
* Comply with all aspects of the treatment, including CT scans, radiographs and 1-year follow-up
* Informed consent

Exclusion Criteria:

* Osteotomy for indication of cartilage treatment or other knee surgeries than unicompartmental OA
* Correction using an open wedge above 10 mm
* Pregnant women at time of enrollment or women who are planning to become pregnant during the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The mean NRS pain score | First week postoperative daily score
  Questionnaire to measure pain.The NRS score is a score between 0 and 10, where 0 means no pain and 10 means the most pain imaginable.

SECONDARY OUTCOMES:
Rehabilitation time | After surgery (+2 weeks, +1 months, +3 months, +6 months, +1 year)
  Time of rehabilitation period (questionnaires)
Reduction of local blood loss | Before surgery and 1 day after surgery
  Amount of blood loss during surgery using haemoglobin measurements
Reduction of local blood loss | Before surgery and a weekly home measurement up to and including 1 month after surgery.
  Amount of blood loss during surgery using calf circumference
Union rate | +1 months, +4 months, +6months, and +12 months
  Bone union determined on xray and CT-scan
Postoperative NRS pain score | After surgery (second week daily score), +1 months, +3months
  Questionnaire to measure pain.The NRS score is a score between 0 and 10, where 0 means no pain and 10 means the most pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: R.J.H. Custers, Dr, Principal Investigator — UMC Utrecht
Locations (1):
- University medical center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Structural allograft impaction enables fast rehabilitation in opening-wedge high tibial osteotomy: a consecutive case series with one year follow-up — https://link.springer.com/article/10.1007/s00167-019-05765-z
- See also: Increasing Fusion Rate Between 1 and 2 Years After Instrumented Posterolateral Spinal Fusion and the Role of Bone Grafting — https://pubmed.ncbi.nlm.nih.gov/32459724/
- See also: Efficacy of a Standalone Microporous Ceramic Versus Autograft in Instrumented Posterolateral Spinal Fusion: A Multicenter, Randomized, Intrapatient Controlled, Noninferiority Trial — https://pubmed.ncbi.nlm.nih.gov/32080013/